CLINICAL TRIAL: NCT05383183
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase IV Trial to Evaluate the Efficacy and Safety of Choline Alfoscerate in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of ChOline ALfoscerate in Patient With Mild to Moderate Alzheimer's Disease
Acronym: COALA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWB-CA400
Record Dates: First submitted 2021-12-06; First posted 2022-05-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline Alfoscerate 1,200mg + Donepezil 5mg or 10mg (Experimental): Oral administration of choline alfoscerate 400mg TID, donepezil QD (evening) for 48 weeks, no dosage change during trial period
  Interventions: Drug: Choline Alfoscerate 400mg
- Placebo + Donepezil 5mg or 10mg (Placebo Comparator): Oral administration of placebo TID, donepezil QD (evening) for 48 weeks, no dosage change during trial period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline Alfoscerate 400mg — Oral administration
  Arms: Choline Alfoscerate 1,200mg + Donepezil 5mg or 10mg
Drug: Placebo — Oral administration
  Arms: Placebo + Donepezil 5mg or 10mg

SUMMARY:
The purpose of this study is to determine whether combination of donepezil, a cholinesterase inhibitor, with choline alfoscerate has a more favourable clinical profile than monotherapy with donepezil alone.

DETAILED DESCRIPTION:
Aging population is a characteristic feature of demographic trends in developed countries. Hence, Alzheimer's disease is recognized as one of today's major healthcare challanges, and its significance will increase even more as the longevity of the population increases. Pre-clinical investigations have suggested that association between ChE-Is (cholinesterase inhibitors) and the cholinergic precursor choline alfoscerate enhances cholinergic neurotransmission more effectively than single compounds alone. This clinical trial is designed to assess if combination of the ChE-I donepezil with choline alfoscerate has a more favorable clinical proﬁle than monotherapy with donepezil alone.

ELIGIBILITY:
Inclusion Criteria:

<Screening Inclusion Criteria>

1. 50 ≤ Age ≤ 85 at time of screening
2. Diagnosed as a probable Alzheimer Dementia patient according to the NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association) criteria
3. 10 ≤ K-MMSE-2 score ≤ 26 at time of screening
4. 0.5 ≤ CDR score ≤ 2 at time of screening
5. Administration of donepezil 5 mg or 10 mg without dose change for at least 3 months at time of screening
6. Ability to walk or to move using a walking aid (i.e. senior walker, cane, or wheelchair)
7. Presence of a caregiver who regularly spends time with the patient and can accompany the patient to hospital visits

   - The caregiver must spend at least 8 hours per week with the patient
   * The caregiver should be able to supervise trial compliance and report subject status to the investigator
8. Sufficient visual acuity, hearing, language ability, motor function and comprehension, as judged by the investigator, to follow the examination procedure (auxiliary devices such as glasses and hearing aids are permitted)
9. Voluntarily decision to participate in this clinical trial from both the subject and the subject's legal representative

<Randomization Inclusion Criteria>

1. 10 ≤ K-MMSE-2 score ≤ 26 at time of randomization
2. Compliance with donepezil ≥ 80% during run-in

Exclusion Criteria:

<Screening Exclusion Criteria>

1. Dementia due to other causes including:

   - Probable vascular dementia according to NINDS-AIREN criteria
   * Infection of the central nervous system (eg HIV, syphilis, etc.)
   * Head trauma
   * Creutzfeld-Jacob disease
   * Pixie's disease
   * Huntington's disease
   * Parkinson's disease
   * Drug addiction and/or Alcoholism
2. Patients with other major structural brain diseases (strategic cerebral infarction, subdural hematoma, traffic hydrocephalus, brain tumor) and/or evidence (CT or MRI results performed within the past 12 months or at screening) as the cause of dementia (provided that (Excluding lacunar cerebral infarction with a diameter of less than 1 cm in the area judged not to be related to cognitive function)
3. 3 ≤ New Rating Scale for ARWMC (Age-Related White Matter Changes) score within 12 months of screening
4. Myocardial infarction, unstable angina pectoris, orthostatic hypotension or unexplained syncope within 12 months of screening, hospitalization for arrhythmia, or moderate to severe congestive heart failure (NYHA class III or IV), clinically Patients with significant structural heart disease (valvular disease, hypertrophic cardiomyopathy)
5. Serious mental disorders such as severe depression, schizophrenia, alcoholism, and drug dependence
6. History of malignant tumor within 5 years of screening. (However, enrollment is allowed if any of the following applies:)

   * More than 5 years since completion of treatment for tumor
   * Basal cell carcinoma, squamous cell carcinoma of the skin, or prostate cancer
7. Genetic problems such as galactose intolerance, lapp lactase deficiency or glucose galactose malabsorption
8. Gastrointestinal diseases (inflammatory bowel disease, etc.) that may affect the absorption of clinical investigational drugs
9. Administration of other dementia treatments (galantamine, rivastigmine, memantine) than donepezil within 3 months of screening
10. Administration of brain function improving drugs (citicoline, oxiracetam, piracetam, choline alfoscerate, Nicergoline, Nimodipine, ginko-biloba, acetyl-l carnitine, etc.) within 1 month of screening
11. Administration of dementia treatments, brain function improving agents, central nervous system stimulants, anticholinergics, tricyclic antidepressants, classic antipsychotics, and hypnotics (excluding short-acting hypnotics) other than experimental drugs during trial period
12. Administration of atypical antipsychotics, anxiolytics, antidepressants (except tricyclic antidepressants), thyroid hormones, short-acting hypnotics, hormone replacement therapy, vitamin E, vitamin B12 supplements, antiparkinsonian drugs, and cholinergic drugs during trial period (However, enrollment is allowed if all of the following apply:)

    - Administration without any changes in dosage within 2 months of randomization

    - Administration without any changes in dosage during trial period

    - except for PRN drugs
13. Hypersensitivity to clinical investigational drugs (choline alfoscerate, donepezil), its components, or piperidine derivatives
14. Possibility of dementia due to abnormalities in vitamin B12, folic acid, and thyroid stimulating hormone (TSH) levels
15. Abnormalities in blood tests at screening:

    - Liver dysfunction: AST or ALT ≥ 3 times the upper limit of normal range

    - Renal dysfunction: Creatinine clearance* < 25 mL/min/1.73 m2

    *MDRD Formula Creatinine clearance (mL/min/1.73m2)= 175 × {serum Creatinine (mg/dL)}- 1.154 × (Age)-0.203 × 0.742 (for female only)
16. Uncontrolled hypertension (SBP>180 mmHg)
17. Illitera
18. Pregnancy and lactation
19. In case of a woman, a patient who does not fall under any of the following:

    * Menopause for at least 2 years at time of screening
    * Contraceptive through surgical methods
20. Deemed inappropriate for enrollment by the investigator for other reasons <Randomization Exclusion Criteria>

1) Abnormalities in blood tests at time of randomization

* Liver dysfunction: AST or ALT ≥ 3 times the upper limit of normal range
* Renal dysfunction: Creatinine clearance* < 25 mL/min/1.73 m2 *MDRD Formula Creatinine clearance (mL/min/1.73m2)= 175 × {serum Creatinine (mg/dL)}- 1.154 × (Age)-0.203 × 0.742 (for female only) 2) Uncontrolled hypertension (SBP>180 mmHg) at the time of randomization 3) Administration of other investigational drugs within the past 3 months from the time of randomization 4) Deemed inappropriate for enrollment by the investigator for other reasons

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Changes in ADAS-Cog scores | 48 weeks from baseline
  ADAS-cog change at 12 and 24 weeks from baseline
  Changes in ADAS-Cog scores at 48 weeks from baseline

SECONDARY OUTCOMES:
Changes in ADAS-Cog scores | Time Frame: 12, 24 weeks from baseline
  Changes in ADAS-Cog scores at 12, 24 weeks from baseline
Changes in ADCOMS scores | 12, 24, and 48 weeks from baseline
  Changes in ADCOMS scores at 12, 24 and 48 weeks from baseline
Changes in K-IADL scores | 12, 24, and 48 weeks from baseline
  Changes in K-IADL scores at 12, 24 and 48 weeks from baseline
Changes in CDR-SB scores | 12, 24, and 48 weeks from baseline
  Changes in CDR-SB scores at 12, 24 and 48 weeks from baseline
Changes in K-MMSE-2 scores | 12, 24, and 48 weeks from baseline
  Changes in K-MMSE-2 scores at 12, 24 and 48 weeks from baseline

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Changwon Fatima Hospital, Changwon
  - Gachon University Gil Medical Center, Incheon
  - CHA Bundang Medical Center, Seongnam
  - The Catholic University of Korea Seoul ST.MARY'S Hospital, Seoul